CLINICAL TRIAL: NCT05578560
Title: Is 3D Optokinetic Stimulation in Virtual Reality Space an Efficient Tool for Improvement of Central Compensation in Patients After Vestibular Schwannoma Surgery?
Brief Title: The Use of Virtual Reality in Rehabilitation in Patients After Vestibular Schwannoma Surgery.
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Charles University, Czech Republic (Other)
Responsible Party: Principal Investigator, Marketa Bonaventurova, Principle investigator, Charles University, Czech Republic
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CharlesU
Record Dates: First submitted 2022-09-16; First posted 2022-10-13 (Actual); Last update posted 2025-06-17 (Actual); Status verified 2025-06

CONDITIONS: Acute Peripheral Vestibulopathy Following Surgical Procedure

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Prehabituation group (Experimental): Patients with vestibular Schwannoma are indicated for the surgery. The patients in this group undergo chemical labyrinthectomy via intratympanically installed gentamicin before the vestibular Schwannoma resection. After the operation, vestibular training under supervision will be performed.
  Interventions: Procedure: Prehabituation; Procedure: Vestibular training
- Virtual reality group (Experimental): Patients with vestibular Schwannoma are indicated for the surgery. After the surgery, they will perform vestibular training under supervision and in addition to this, they will be exposed to 3D optokinetic stimulation in virtual reality space.
  Interventions: Procedure: 3D optokinetic stimulation in virtual reality space; Procedure: Vestibular training
- Vestibular training group (Experimental): Patients with vestibular Schwannoma are indicated for the surgery. After the surgery, they will perform vestibular training under supervision.
  Interventions: Procedure: Vestibular training

INTERVENTIONS:
Procedure: Prehabituation — chemical labyrinthectomy with intratympanically installed gentamicin
  Arms: Prehabituation group
Procedure: 3D optokinetic stimulation in virtual reality space — 3D optokinetic stimulation via virtual reality goggles with the software designed by Pro-Zeta comp.
  Arms: Virtual reality group
Procedure: Vestibular training — vestibular training program adopted for patients with acute vestibular loss under the supervision of a physical therapist. The program includes gaze stability exercises, smooth pursuit, and saccadic eye movements, and postural exercises to improve balance control and gait stability. Each session lasts around 30 minutes and happened daily for the 7 postoperative days.

SUMMARY:
Resection of the vestibular schwannoma leads to acute peripheral or combined vestibular loss caused by a surgical lesion to the branches of the vestibular nerve and, less frequently also the lesion of the cerebellum. The lesion presents in patients with postural instability, vertigo, oscillopsia, and vegetative symptoms that may accompany it. The organism reacts to this state with the process of central compensation with the significant role of the cerebellum. The goal of the rehabilitation is to support this process and thus to make recovery faster and more efficient since not all patients are capable of complete restoration of the vestibular function. Up to date, rehabilitation includes, apart from the specific vestibular exercise, also the possibility of modern techniques using virtual reality space and prehabituation. Thanks to prehabituation, i.e., chemical labyrinthectomy with intratympanically installed gentamicin, the timing of the origin of the acute vestibular loss and the surgical procedure is separated. Therefore, there is a chance of achieving vestibular compensation before vestibular schwannoma removal. In the last decade, due to the advances in technology in the field of computer games and the applications for smartphones, the tools for virtual reality have become less expensive and more available in common praxis. Virtual reality is a technique for generating an environment that can strengthen three-dimensional optokinetic stimulation, subsequently the process of central compensation. Overall, it may shorten the time of recovery after the surgery and improve patients' quality of life.

DETAILED DESCRIPTION:
This study was approved by institutional ethics committee of the University Hospital Motol and all patients provide inform consent prior to study commencement.

In this prospective randomized single-center study, we will enroll patients who undergo vestibular schwannoma resection in our department. All patients must be found to be indicated for the surgery. The size of the tumor will be classified according to the Koos classification. The patients with hearing loss will undergo prehabituation (group A). The rest of the patients will be randomly divided into either a virtual reality group (group B), or the control group (group C). Two days before the surgery (time 1) all of the patients will undergo a clinical oto-neurological examination as well as examination by objective methods - video-nystagmography (VNG), air calorics, video Head Impulse Test (vHIT), and cervical Vestibular Evoked Myogenic Potentials (cVEMP). They will also fill out a set of questionnaires - the Penn Acoustic Neuroma Quality-Of-Life scale (PANQOL), Dizziness Handicap Inventory (DHI), Generalized Anxiety Disorder 7 - item scale (GAD-7), and Self-rating Depression Scale (SDS). All of them were translated into the Czech language. In addition to it, we used the in-house questionnaire focused on vertigo symptoms.

On the second day after the surgery, all groups of patients begin to practice the vestibular training program adopted for patients with acute vestibular loss under the supervision of a physical therapist. The program includes gaze stability exercises, smooth pursuit, and saccadic eye movements, and postural exercises to improve balance control and gait stability. Each session will last around 30 minutes and will happen daily for the whole time of the hospitalization, thus seven days. Additionally, during that time, group B will obtain seven sessions of 30-minute-long optokinetic stimulation via virtual reality goggles. Subjective and objective assessments will be repeated at the hospital discharge which is on the 7-10th postoperative day (time 2) and 3 months after surgery (time 3).

ELIGIBILITY:
Inclusion Criteria:

* Vestibular Schwannoma appropriate to surgical resection

Exclusion Criteria:

* Eye disorder
* Oculomotor disorder in patient history
* Nerve palsy other than n. VIII, n. VII.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2020-01-01 (Actual); Primary Completion 2026-06 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
video Head Impulse Test | 10 days after the surgery
  Objective method. The video head impulse test is an ear-specific test that detects disorders of the vestibulo-ocular reflex and identifies which ear is affected in cases of peripheral vestibular loss. It can test all three semicircular canal in each ear independently. Patients with a vestibular loss exhibit a corrective saccadic eye movement (a "catch-up" saccade) either during or after the head impulse and the gain of the head in comparison to the eye will not be equivalent.
video Head Impulse Test | 3 months after the surgery
  Objective method. The video head impulse test is an ear-specific test that detects disorders of the vestibulo-ocular reflex and identifies which ear is affected in cases of peripheral vestibular loss. It can test all three semicircular canal in each ear independently. Patients with a vestibular loss exhibit a corrective saccadic eye movement (a "catch-up" saccade) either during or after the head impulse and the gain of the head in comparison to the eye will not be equivalent.
Vestibular evoked myogenic potentials | 10 days after the surgery
  Objective method. Vestibular evoked myogenic potentials are short-latency, vestibular-dependent reflexes that are recorded from the sternocleidomastoid muscles in the anterior neck (cervical VEMPs - cVEMPs) and the inferior oblique extraocular muscles (ocular VEMPs - oVEMPs). They are evoked by short bursts of sound delivered through headphones (air conducted) or vibration applied to the skull (bone conducted). As these stimuli have been shown to preferentially activate otolith organs rather than semicircular canals, VEMPs are used clinically as measures of otolith function. They are used to reveal loss of otolith function, i.e. in conditions where damage to the inner ear, vestibular nerve, or central vestibular pathways occurs.
Vestibular evoked myogenic potentials | 3 months after the surgery
  Objective method. Vestibular evoked myogenic potentials are short-latency, vestibular-dependent reflexes that are recorded from the sternocleidomastoid muscles in the anterior neck (cervical VEMPs - cVEMPs) and the inferior oblique extraocular muscles (ocular VEMPs - oVEMPs). They are evoked by short bursts of sound delivered through headphones (air conducted) or vibration applied to the skull (bone conducted). As these stimuli have been shown to preferentially activate otolith organs rather than semicircular canals, VEMPs are used clinically as measures of otolith function. They are used to reveal loss of otolith function, i.e. in conditions where damage to the inner ear, vestibular nerve, or central vestibular pathways occurs.
Videonystagmography | 10 days after the surgery
  Objective method. It is a technology for testing inner ear and central motor functions, a process known as vestibular assessment. It involves the use of infrared goggles to trace eye movements during visual stimulation and positional changes.
Videonystagmography | 3 months after the surgery
  Objective method. It is a technology for testing inner ear and central motor functions, a process known as vestibular assessment. It involves the use of infrared goggles to trace eye movements during visual stimulation and positional changes.
Dizzines Handicap Inventory | 10 days after the surgery
  Subjective method. It evaluates the self-perceived handicapping effects of dizziness in everyday life imposed by vestibular system disease. It contains 25-items, which are subgrouped into three content domains representing functional, emotional and physical aspects of dizziness and unsteadiness. Scoring of the DHI is as follows, a "yes" answer is awarded 4 points, "sometimes," 2 points and "no," 0 points. Possible scores range from 0, suggesting no handicap, to 100, indicating significant self-perceived handicap.
Dizzines Handicap Inventory | 3 months after the surgery
  Subjective method. It evaluates the self-perceived handicapping effects of dizziness in everyday life imposed by vestibular system disease. It contains 25-items, which are subgrouped into three content domains representing functional, emotional and physical aspects of dizziness and unsteadiness. Scoring of the DHI is as follows, a "yes" answer is awarded 4 points, "sometimes," 2 points and "no," 0 points. Possible scores range from 0, suggesting no handicap, to 100, indicating significant self-perceived handicap.
Generalized Anxiety Disorder - 7item scale | 10 days after the surgery
  Subjective method. This questionnaire is a valid and efficient tool for screening for generalized anxiety disorder and assessing its severity in clinical practice and research. Because of the 7 items is scored from 0 to 3, the GAD- 7 scale score ranges from 0 to 21. Increasing scores on the scale are strongly associated with the functional impairment.
Generalized Anxiety Disorder - 7item scale | 3 months after the surgery
  Subjective method. This questionnaire is a valid and efficient tool for screening for generalized anxiety disorder and assessing its severity in clinical practice and research. Because of the 7 items is scored from 0 to 3, the GAD- 7 scale score ranges from 0 to 21. Increasing scores on the scale are strongly associated with the functional impairment.
Penn Acoustic Neuroma Quality-Of-Life scale | 10 days after the surgery
  Subjective method. This questionnaire is a valid and reliable disease-specific quality of life instrument for acoustic neuroma. Since the vestibular schwannomas are benign tumors such quality of life is a paramount of importance when considering treatment options. It consists of 26 questions covering all relevant domains such as hearing, balance, anxiety, energy, pain and general. Answer to each question is scored in range from 1 to 5, meaning the total score ranges from 26 to 130, the higher score indicates the worse quality of life.
Penn Acoustic Neuroma Quality-Of-Life scale | 3 months after the surgery
  Subjective method. This questionnaire is a valid and reliable disease-specific quality of life instrument for acoustic neuroma. Since the vestibular schwannomas are benign tumors such quality of life is a paramount of importance when considering treatment options. It consists of 26 questions covering all relevant domains such as hearing, balance, anxiety, energy, pain and general. Answer to each question is scored in range from 1 to 5, meaning the total score ranges from 26 to 130, the higher score indicates the worse quality of life.
Self-rating Depression Scale | 10 days after the surgery
  Subjective method. It assess depression simply and specifically as a psychiatric disorder. It is constructed so that the less depressed patient and his complaints will have low score on the scale, and the more depressed patient and his complaints will have a higher score. In scoring SDS, which contains 20 items, a value of 1 to 4 is assigned to a response depending upon whether the item was worded positively or negatively. An index for the SDS was derived by dividing the sum of the values obtained on the 20 items by the maximum possible score of 80 and expressed as a decimal.
Self-rating Depression Scale | 3 months after the surgery
  Subjective method. It assess depression simply and specifically as a psychiatric disorder. It is constructed so that the less depressed patient and his complaints will have low score on the scale, and the more depressed patient and his complaints will have a higher score. In scoring SDS, which contains 20 items, a value of 1 to 4 is assigned to a response depending upon whether the item was worded positively or negatively. An index for the SDS was derived by dividing the sum of the values obtained on the 20 items by the maximum possible score of 80 and expressed as a decimal.

CONTACTS AND LOCATIONS:
Overall Officials: Markéta Bonaventurová, Principal Investigator — Department of ENT and Head and Neck Surgery, Charles University in Prague and Motol University Hospital
Locations (1):
- Department of Otorhinolaryngology and Head and Neck Surgery, 1st Faculty of Medicine Charles University and Motol University Hospital, Postgraduate Medical School, Prague, Czechia

REFERENCES:
- [Background] Balatkova Z, Cada Z, Hruba S, Komarc M, Cerny R. Assessment of visual sensation, psychiatric profile and quality of life following vestibular schwannoma surgery in patients prehabituated by chemical vestibular ablation. Biomed Pap Med Fac Univ Palacky Olomouc Czech Repub. 2020 Dec;164(4):444-453. doi: 10.5507/bp.2019.056. Epub 2019 Dec 3. PMID 31796939
- [Background] Cada Z, Balatkova Z, Chovanec M, Cakrt O, Hruba S, Jerabek J, Zverina E, Profant O, Fik Z, Komarc M, Betka J, Kluh J, Cerny R. Vertigo Perception and Quality of Life in Patients after Surgical Treatment of Vestibular Schwannoma with Pretreatment Prehabituation by Chemical Vestibular Ablation. Biomed Res Int. 2016;2016:6767216. doi: 10.1155/2016/6767216. Epub 2016 Dec 8. PMID 28053986